CLINICAL TRIAL: NCT00314808
Title: A Pilot Study of Dronabinol for Adult Patients With Primary Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007559; 7136-05-6R0 (Other: Duke legacy protocol number)
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Brain Neoplasms; Nausea; Vomiting
Keywords: primary gliomas; brain tumors; vomiting; appetite suppression; appetite
MeSH Terms: conditions — Brain Neoplasms; Nausea; Vomiting | interventions — Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dronabinol (Experimental)
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol — Oral route, 5mg PO 2x daily before and during 2 cycles of chemotherapy,2.5mg PO every night when not on chemotherapy
  Other Names: delta-9-Tetrahydrocannabinol

SUMMARY:
This study seeks to define the tolerability and safety associated with the administration of Dronabinol in the treatment of adults with nausea, vomiting and appetite loss in patients with primary gliomas who are undergoing chemotherapy treatment. The study will also describe the effect of Dronabinol on the quality of life in terms of nausea, vomiting and anorexia in this patient group.

DETAILED DESCRIPTION:
Symptoms identified as impacting quality of life include nausea and vomiting, appetite changes, pain, fatigue, mobility, insomnia, mood, bowel patterns, concentration and appearance (Donaldson and Fields, 1998). There has been little information published on the impact of these symptoms in the glioblastoma multiforme (GBM) population. More specifically, to date, there has not been an investigation that demonstrates the efficacy of an intervention on improving appetite, and decreasing nausea and vomiting in patients with GBM. This need serves as the basis for the current proposed investigation utilizing Dronabinol, a cannabinoid known to decrease incidence of nausea and vomiting, as well as controlling appetite changes for terminally ill patients receiving chemotherapy. In addition, there is no published research on the use of Dronabinol and dose limited toxicity for the brain tumor population.

In this study, patients will receive daily Dronabinol therapy through their chemotherapy cycle. Patients will complete daily appetite and nausea/vomiting logs, as well as receive telephone follow-up from the research coordinator to assess impact of treatment. This will be assessed through two consecutive cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of primary malignant brain tumor (grade 3 or 4)
* Karnofsky greater than or equal to 80%
* Life expectancy greater than or equal to 6 months
* Patients must be undergoing one of the following chemotherapy administrations: Temozolomide; Lomustine (CCNU) or Irinotecan or Camptosar (CPT-11)
* Patients must give written informed consent
* Patients must have aspartate aminotransferase (AST), alanine transaminase (ALT), total serum bilirubin, and alkaline phosphatase less than 2 times upper limits of normal laboratory values, performed within 14 days prior to initiation of study
* For women, negative risk of pregnancy through standard chemotherapy screening procedures inclusive of pregnancy test, menopause or surgical procedure
* Patient must have social support with caregiver daily monitoring for side effects

Exclusion Criteria:

* Premorbid central nervous system (CNS) diagnosis (cerebral vascular accident (CVA), closed head injury (CHI), multiple sclerosis (MS)
* Patients with global aphesis limiting the informed consent process
* Patients with unmanaged psychiatric disease
* Patients with history of drug addiction or recent illicit drug usage within the last 3 months
* Patients with hypersensitivity to dronabinol, marijuana or sesame seed oil
* Patients must not be taking an concomitant meds contraindicated with Dronabinol (including anxiolytics, sedative, hypnotics, barbiturates, general anesthetics, monoamine oxidase inhibitors [MAOIs], opiate agonists, phenothiazines, sedating H1 blockers, skeletal muscle relaxants and sympathomimetics)
* Patients who have hepatic enzyme elevation of greater than two times upper limits of normal laboratory values for AST, ALT, total serum bilirubin or alkaline phosphatase
* Pregnant or breastfeeding women
* Women of childbearing potential who are not using an effective method of contraception (oral contraceptives, female and/or male barrier devices, spermicidal agents, or surgical procedures inhibiting contraception)
* Patients who live alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-04; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah H Allen, MSN, RN, CNS, FNP-BC, AOCNP, Principal Investigator — Duke University
Locations (1):
- Preston Robert Tisch Brain Tumor Center at Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were accrued between May 2006 and June 2009 within the clinic at Duke Comprehensive Cancer Center.
Groups:
- Dronabinol: Dronabinol 5 mg BID administered 24 hours prior to, during, and 48 hours after completion of oral/intravenous chemotherapy for a maximum of 2 consecutive cycles
Period: Overall Study
Arm/Group | Dronabinol
Started | 33
Completed | 25 (Completed 2 cycles of Dronabinol or terminated early due to treatment-related adverse events (AE))
Not Completed | 8
Not completed — Disease Progression without AE | 4
Not completed — Withdrawal by Subject/PI without AE | 4

BASELINE CHARACTERISTICS:
Arm/Group | Dronabinol
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Tolerability Rate
Description: Percentage of participants where the 2 cycles of Dronabinol is tolerable. The treatment regimen is considered intolerable if (1) at least two adverse events of the following types that are attributed to Dronabinol during the 2 cycles of treatment occur: ≥Grade 3 non-hematologic, ≥Grade 2 hepatic/metabolic or ≥Grade 4 neuro toxicities, or (2) Dronabinol treatment is terminated early due to adverse events
Time Frame: Two months
Population: 25 of the 33 patients treated with Dronabinol completed 2 cycles of protocol treatment or terminated protocol treatment due to adverse events. The remaining 8 patients are excluded from this tabulation as they terminated Dronabinol treatment before completion of 2 cycles of treatment for reasons unrelated to adverse events.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dronabinol
Number analyzed (Participants) | 25
percentage of participants | 60 [39 to 79]

2. Primary Outcome: Unacceptable Toxicity Rate
Description: Percentage of participants who experience one or more adverse events attributable to Dronabinol of the following types or grades: ≥Grade 3 non-hematologic, ≥Grade 2 hepatic/metabolic or ≥Grade 4 neuro toxicities
Time Frame: 2 months
Population: All treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dronabinol
Number analyzed (Participants) | 33
percentage of participants | 0 [0 to 11]

3. Secondary Outcome: Mean Change From Baseline in Quality of Life -- FACT-Br
Description: The mean change between baseline and post-treatment in quality of life as measured by the Functional Assessment of Cancer Therapy-Brain (FACT-Br), where change is computed as quality of life at 2 months minus quality of life at baseline. The FACT-Br instrument consists of 54 items to assess physical(PWB), social and family (SWB), emotional (EWB), functional well-being (FWB), and additional brain cancer specific concerns (AC). Using a 5-point Likert type scale, responses to individual items range from 0 (not at all) to 4 (Very Much) with higher scores indicating better quality of life. PWB, SWB, and FWB are the sum of 7 items and have a possible range between 0 and 28. EWB ranges between 0 and 24, and is the sum of 6 items. AC is the sum of 19 items, and ranges between 0 and 76.
Time Frame: baseline and 2 months
Population: 19 patients provided both baseline and follow-up assessments; however, only 11 patients provided adequate information to compute the score for the additional brain cancer specific concerns subscale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dronabinol
Number analyzed (Participants) | 19
units on a scale
  Physical Well-Being (N=19) | 1.68 (6.75)
  Social Well-Being (N=19) | 0.47 (3.58)
  Emotional Well-Being (N=19) | 1.58 (6.1)
  Functional Well-Being (N=19) | 2.26 (6.33)
  Additional Concerns (N=11) | 1.77 (11.2)

4. Secondary Outcome: Mean Change From Baseline in Quality of Life -- FLIE
Description: The mean change from baseline in quality of life as measured by the Functional Living Index Emesis (FLIE) scale during the first 24 and 72 hours of cycle 1. Change at 24 hours was computed as the 24 hour FLIE assessment minus the baseline assessment; whereas, change at 72 hours was computed as the 72 hour FLIE assessment minus the baseline assessment. The FLIE consists of 18 items for nausea and appetite on a 7-point scale. The effect of nausea and vomiting is measured by physical activity, social, and emotional function. Higher scores indicate less difficulty and interference with nausea and vomiting. Scores for the two subscales (nausea and vomiting) range between 0 and 54.
Time Frame: baseline, 24 hours, and 72 hours
Population: For cycle 1, 28 patients with a baseline and follow-up assessment are included in the analysis of change at 24 and 72 hours.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dronabinol
Number analyzed (Participants) | 28
units on a scale
  Nausea at 24 hours | -13.07 (3.50)
  Nausea at 72 hours | -4.18 (3.52)
  Emesis at 24 hours | -10.96 (3.10)
  Emesis at 72 hours | -3.50 (2.82)

5. Secondary Outcome: Mean Change From Baseline in Quality of Life -- MMSE
Description: The mean change between baseline and post-treatment in quality of life as measured by the Mini Mental Status Exam (MMSE). Change is computed as the MMSE level at month 2 minus MMSE level at baseline. MMSE is an 11-item questionnaire used to measure global cognitive status with scores ranging from 0 to 30; higher scores are an indication of greater cognitive function.
Time Frame: baseline and 2 months
Population: 17 patients provided both a pre- and post-treatment assessment of MMSE.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dronabinol
Number analyzed (Participants) | 17
units on a scale | 1.41 (3.47)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Dronabinol
Serious Adverse Events (participants affected / at risk) | 1/33
Other Adverse Events (participants affected / at risk) | 12/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dronabinol (N=33)
Wound infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dronabinol (N=33)
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 2
Cognitive disturbance (Nervous system disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 4
Dysphasia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No